CLINICAL TRIAL: NCT01284751
Title: The Use of Major Depression Inventory (MDI) in Measuring Preoperative Depressive Symptoms in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: M.D. Melissa Voigt Hansen, Herlev Hospital - Department of surgical gastroenterology
Other Study IDs: MVH-04; H-1-2010-FSP (Other: The Danish Ethics Committee)
Record Dates: First submitted 2011-01-24; First posted 2011-01-27 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Depression; Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients: Patients aged 30-70 years having a lumpectomy or mastectomy at the Department of Breast Surgery at Herlev Hospital, Copenhagen, Denmark.
  Interventions: Other: MDI - self-rating inventory

INTERVENTIONS:
Other: MDI - self-rating inventory — MDI with 12 questions to be completed approximately 1 week before surgery

SUMMARY:
The purpose of this study is to measure depressive symptoms in breast cancer patients before surgery with Major Depression Inventory (MDI). The investigators hypothesize that this patient group will not produce scores correlating to having a mild, moderate or severe depression even though they have just recently experienced a major life crisis by receiving a malignant diagnosis.

DETAILED DESCRIPTION:
The Major Depression Inventory is a self-rating depression scale with 12 questions. The questionnaire has previously been investigated in a Danish population. The scale contains the 10 ICD-10 (International Classification of Diseases)symptoms of depression and these symptoms are identical with the DSM-IV major depression symptoms with the exception of one symptom, low self-esteem, which in DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) is incorporated in the symptom of guilt. On a six-point Likert scale, the individual items measure how much of the time the symptoms have been present during the last 14 days. The MDI is then scored according to specific guidelines and can be used as both a rating scale and a diagnostic instrument.

Patients will approximately one week after the diagnosis of breast cancer has been made, corresponding to approximately one week before surgery, be asked to complete the MDI. Patients therefore only complete the MDI once in the whole study. At the same time a Mini Mental State Examination (MMSE) and questions regarding previous illnesses and medication will be asked. Patients will not be followed up in any way.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-70 years old, who are undergoing a lumpectomy or mastectomy
* ASA I-III

Exclusion Criteria:

* Planned or ongoing preoperative chemotherapy
* Known and treated sleep apnea syndrome
* Insulin treated diabetes mellitus
* Known or previous treated depressive illness or bipolar disorder
* Known autoimmune disease
* Incompensated cirrhosis
* Other previous or ongoing cancer
* Known medically treated sleep disorder (insomnia, restless legs etc)
* Shift-work or night-work
* Daily alcohol intake of more than 5 units
* Preoperative treatment with psychopharmacological drugs, opioids or anxiolytics
* Predicted bad compliance
* Pregnant or breast feeding
* Preoperative MMSE score less than 24

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Breast Surgery
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Approximately one week before surgery
  Total score on the Major Depression Inventory. When used as a diagnostic instruemtn patients witll according to the ICD-10 algorhythym be classified as mild, moderate or severe depression or no depression.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa V Hansen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Background] Olsen LR, Jensen DV, Noerholm V, Martiny K, Bech P. The internal and external validity of the Major Depression Inventory in measuring severity of depressive states. Psychol Med. 2003 Feb;33(2):351-6. doi: 10.1017/s0033291702006724. PMID 12622314
- [Background] Bech P, Rasmussen NA, Olsen LR, Noerholm V, Abildgaard W. The sensitivity and specificity of the Major Depression Inventory, using the Present State Examination as the index of diagnostic validity. J Affect Disord. 2001 Oct;66(2-3):159-64. doi: 10.1016/s0165-0327(00)00309-8. PMID 11578668
- [Background] Olsen LR, Mortensen EL, Bech P. Prevalence of major depression and stress indicators in the Danish general population. Acta Psychiatr Scand. 2004 Feb;109(2):96-103. doi: 10.1046/j.0001-690x.2003.00231.x. PMID 14725589